CLINICAL TRIAL: NCT06204354
Title: Construction of Gynecological Tumor Sample Library
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Construction of tumor sample
Record Dates: First submitted 2023-12-22; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-12

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh samples from gynecological cancer, including cervical cancer, ovarian cancer, endometrial cancer, vulva cancer, vaginal cancer, and some other rare type of cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- samples of cervical cancer: fresh samples collected from patients diagnosed with cervical cancer
- samples of endometrial cancer: fresh samples collected from patients diagnosed with endometrial cancer
- samples of ovarian cancer: fresh samples collected from patients diagnosed with ovarian cancer
- samples of vulva cancer: fresh samples collected from patients diagnosed with vulva cancer
- samples of vaginal cancer: fresh samples collected from patients diagnosed with vaginal cancer
- samples of rare gynecological cancer: fresh samples collected from patients diagnosed with rare gynecological cancer

SUMMARY:
Constructing a gynecological tumor samples library, which is open and can be accessed.

DETAILED DESCRIPTION:
This project is the construction and maintenance of a gynecological tumor sample library. It is supported by the National Key Laboratory of Difficult, Severe, and Rare Diseases at Peking Union Medical College Hospital of the Chinese Academy of Medical Sciences. This project will lay a clinical specimen foundation for exploring the molecular mechanisms of gynecological tumors in the future.

ELIGIBILITY:
Inclusion Criteria:

1. An informed consent form was obtained. If the age is less than 18 years old, the consent form should be signed by the guardian.
2. Preoperative tumor burden assessment and intraoperative evaluation by the supervising physician (professor) suggest sampling is acceptable.
3. The research team believes that sampling is possible.
4. Having the relevant requirements for sample library storage.
5. Surgical treatment is performed at Peking Union Medical College Hospital.

Exclusion Criteria:

1. Not meeting all inclusion criteria.
2. The research team considers any circumstances or considerations that may hinder normal pathological evaluation.

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with gynecologic cancer, including cervical cancer, endometrial cancer, ovarian cancer, vulva cancer, vaginal cancer, and other rare type gynecologic cancer.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
construction of Biobank | 3 years
  Biobank including gynecolgic cancer samples, including cervical cancer, endometrial cancer, ovarian cancer, vulva cancer, vaginal cancer, and others types

SECONDARY OUTCOMES:
Exploring the molecular mechanism based on biobank | 3 year
  Exploring the molecular mechanism of gynecological tumor pathogenesis based on biobank
Drug sensitivity detection based on biobank | 3 year
  Exploring drug sensitivity detection in gynecological tumors based on biobank